CLINICAL TRIAL: NCT04130815
Title: Effect of Aerosol Particle Size and Breathing Pattern of Inhalation on Relief of Experimentally Induced Air Hunger by Inhaled Furosemide
Brief Title: Aerosol Particle Size and Breathing Pattern During Inhaled Furosemide
Acronym: FurAH-II
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr. Shakeeb H Moosavi, Senior Lecturer in Clinical Physiology, Oxford Brookes University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: L19185
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: Furosemide will be inhaled on 4 separate days each with a different pattern of breathing/droplet size combination. The four combinations will be: (i) slow/deep breathing with small droplet size, (ii) slow/deep breathing with large droplet size, (iii) fast/shallow breathing with large droplet size and (iv) fast/shallow breathing with small droplet size.
Who Masked: Participant
Masking Description: Participants will not know which droplet size they will be receiving on any one test day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Slow/Deep/Large (Active Comparator): Slow/deep breathing pattern will be targeted while inhaling furosemide with nebulizer set to deliver 4ml of a 10mg/ml solution of furosemide with large droplet size over a 10-15 minute duration
  Interventions: Drug: Inhaled furosemide
- Slow/Deep/Small (Active Comparator): Slow/deep breathing pattern will be targeted while inhaling furosemide with nebulizer set to deliver 4ml of a 10mg/ml solution of furosemide with small droplet size over a 10-15 minute duration.
  Interventions: Drug: Inhaled furosemide
- Fast/Shallow/Large (Active Comparator): Fast/shallow breathing pattern will be targeted while inhaling furosemide with nebulizer set to deliver 4ml of a 10mg/ml solution of furosemide with large droplet size over a 10-15 minute duration.
  Interventions: Drug: Inhaled furosemide
- Fast/Shallow/Small (Active Comparator): Fast/shallow breathing pattern will be targeted while inhaling furosemide with nebulizer set to deliver 4ml of a 10mg/ml solution of furosemide with small droplet size over a 10-15 minute duration.
  Interventions: Drug: Inhaled furosemide

INTERVENTIONS:
Drug: Inhaled furosemide — 4ml of 10mg/ml solution of furosemide nebulized with small and large droplet sizes and inhaled with different breathing patterns
  Other Names: Lasix

SUMMARY:
The study hypothesises that the variability in relief of air hunger with inhaled furosemide that is reported in previous studies can be explained by the breathing pattern adopted during the inhalation and the droplet size in the aerosol, both of which would influence the site of deposition of the aerosol in the lungs

DETAILED DESCRIPTION:
Recent studies suggest that inhaling furosemide as a mist reduces air hunger in healthy volunteers in whom air hunger is induced experimentally in the lab. However, how much reduction varies among individuals. It is not known if the way the mist is breathed (slow/deep or fast/shallow) or the size of the droplets in the mist (large or small) can explain the variation in relief. Both of these factors can influence the site of deposition of the aerosol in the lungs

In this study the relief of air hunger (induced by hypercapnia and constrained ventilation) will be compared when furosemide is inhaled quickly or slowly, and when the mist has large or small droplets. 20 healthy volunteers will be recruited. After a practice session, the 'air hunger' test will be performed before and after 4ml of a 10mg/ml solution of furosemide (40mg). This will be repeated on 4 separate test days using a different method of inhaling the furosemide on each day.

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers aged 18 and over

Exclusion Criteria:

* On any medication, including herbal medication (other than mild analgesics, vitamins and mineral supplements or, for females, oral contraceptives), whether prescribed or over-the-counter, in the two weeks prior to test sessions involving administration of furosemide or saline.
* Female participants who are pregnant, lactating or planning pregnancy over the course of trial
* A medical history of heart, kidney or liver disease/electrolyte disturbances/ immunosuppression/frequent fainting episodes/COPD/nasal polyps/Addison's/acute porphyria/significant prostatic symptoms/acute gout attack/life expectancy <6months or history of allergic reaction to furosemide and/or any of the other ingredients of furosemide or amiloride, sulfonamides or sulphonamide derivatives, such as sulfadiazine or co-trimoxazole
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Have participated in another research trial involving an investigational product in the past 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for air hunger | Final minute of a 5 minute steady state period per breathing test
  The visual analogue scale (VAS) is from 0 (no air hunger) to 100 (extreme air hunger -tolerable limit). The VAS ratings are taken every 15 seconds during each experimentally induced air hunger test. Each breathing test (hypercapnia with constrained ventilation) is performed before and after each mist inhalation. The final minute of a 5 minute steady state period of hypercapnia and constrained ventilation is analysed during each breathing test (8 breathing tests in total)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grogono JC, Butler C, Izadi H, Moosavi SH. Inhaled furosemide for relief of air hunger versus sense of breathing effort: a randomized controlled trial. Respir Res. 2018 Sep 20;19(1):181. doi: 10.1186/s12931-018-0886-9. PMID 30236110